CLINICAL TRIAL: NCT05428410
Title: Study on Biomarkers to Predict the Efficacy of IL-4R Monoclonal Antibody（CM310） for Chronic Rhino-sinusitis With Polyps
Brief Title: Study on Biomarkers to Predict the Efficacy of IL-4R Monoclonal Antibody for Chronic Rhino-sinusitis With Polyps
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TR-CM310 treatment biomarker
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-05

CONDITIONS: Chronic Rhino-sinusitis; IL-4R; Monoclonal Antibody; Biomarker

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Polyps of chronic rhino-sinusitis with polyps
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IL-4R responders: IL-4R was injected subcutaneously. Base line and treatment end point nasal polyp score were compared and NPS >1.
  Interventions: Other: IL-4R
- IL-4R nonresponders: IL-4R was injected subcutaneously. Base line and treatment end point nasal polyp score were compared and NPS ≤1.
  Interventions: Other: IL-4R
- Controls: Placebo was injected subcutaneously.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: IL-4R — IL-4R was injected subcutaneously.
  Groups: IL-4R nonresponders; IL-4R responders
Other: Placebo — Placebo was injected subcutaneously.
  Groups: Controls

SUMMARY:
The prevalence of chronic rhinosinusitis in China is about 8%, and some patients still suffer from recurrences after surgery and drug treatment. Monoclonal antibody is considered to be a new drug strategy that can significantly improve the control rate of such patients, but there is a lack of markers to guide the selection of monoclonal antibodies. The price of monoclonal antibody is expensive, which calls for screening markers for predicting the efficacy of monoclonal antibody and precisely implementing this treatment strategy. In addition, it can also improve the quality of life of patients and reduce the social and economic burden.

Beijing Tongren Hospital, Capital Medical University recently completed a randomized, double-blind, placebo-controlled, phase II clinical study which included multiple subcutaneous administration of CM310 recombinant humanized monoclonal antibody injection in patients with chronic sinusitis and nasal polyps to evaluate the efficacy and safety as well as the pharmacokinetics, pharmacodynamics, immunogenicity and preliminary efficacy(NCT04805398). The therapeutic target of CM310 recombinant humanized monoclonal antibody injection is IL-4R. The unblinded data showed significant differences in the efficacy of the subjects and we started the investigator-initiate trial (IIT) study aiming at investigating the remaining samples of the project and carrying out a biomarker study to screen and predict the efficacy of IL-4R monoclonal antibody.

DETAILED DESCRIPTION:
The prevalence of chronic rhinosinusitis in China is about 8%, and some patients still suffer from recurrences after surgery and drug treatment. Monoclonal antibody is considered to be a new drug strategy that can significantly improve the control rate of such patients, but there is a lack of markers to guide the selection of monoclonal antibodies. The price of monoclonal antibody is expensive, which calls for screening markers for predicting the efficacy of monoclonal antibody and precisely implementing this treatment strategy. In addition, it can also improve the quality of life of patients and reduce the social and economic burden.

Beijing Tongren Hospital, Capital Medical University recently completed a randomized, double-blind, placebo-controlled, phase II clinical study which included multiple subcutaneous administration of CM310 recombinant humanized monoclonal antibody injection in patients with chronic sinusitis and nasal polyps to evaluate the efficacy and safety as well as the pharmacokinetics, pharmacodynamics, immunogenicity and preliminary efficacy(NCT04805398, detailed in https://clinicaltrials.gov/ct2/show/NCT04805398). The therapeutic target of CM310 recombinant humanized monoclonal antibody injection is IL-4R. The unblinded data showed significant differences in the efficacy of the subjects and we started the IIT study aiming at investigating the remaining samples of the project and carrying out a biomarker study to screen and predict the efficacy of IL-4R monoclonal antibody.

The biomarker levels between IL-4R responders(Defined as Nasal Polyps Score (NPS)>1 at 16 months after subcutaneously CM310) and IL-4R nonresponders (Defined as Nasal NPS≤1 at 16 months after subcutaneously CM310)were compared. The biomarker levels between IL-4R and control groups were also compared.

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled in NCT04805398.

Exclusion Criteria:

Patients not enrolled in NCT04805398.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients wih Bilateral CRSwNP. Prior treatment with systemic corticosteroids (SCS), and/or contraindicate to or intolerance to SCS, and/or with prior surgery to nasal polyps.
  Stable dose of intranasal corticosteroids for at least 4 weeks before screening. Ongoing symptoms for at least 4 weeks before screening as ptients enrolled in NCT04805398.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2022-06-17 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Base line sirius red staining and immunopathological staining | Base line
  Base line sirius red staining and immunopathological staining
End point sirius red staining and immunopathological staining | at Week 16
  End point sirius red staining and immunopathological staining

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Study Chair — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
We haven't decided sharing the IPD yet.